CLINICAL TRIAL: NCT02138071
Title: Psychological Variables in Physiotherapy Treatment for LBP: a Comparison Between Individual and Gruop Treatment
Brief Title: Psychological Variables in Physiotherapy Treatment of Low Back Pain: A Comparison of Group and Individual Treatment
Status: Completed | Type: Observational
Sponsor: Bait Balev Hospital (Other)
Collaborators: Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor
Other Study IDs: 12/2012; NCT01640132 (obsolete NCT alias)
Record Dates: First submitted 2014-05-13; First posted 2014-05-14 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2015-06

CONDITIONS: Low Back Pain
Keywords: low back pain; lumbar pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Individual: Treatment in the 'Individual group therapy' will include physiotherapy protocols usually used by physiotherapist working at Maccabi Healthcare Services (Exercises, Modalities, Maual therapy and Back Care education)
- group: Participants in group therapy will receive 6-8 group treatments (6-12 pateints per group) which will also include exercises and back-care education. No intervention will be done by the investigator.Therapists will use protocols commonly used in Maccabi Healthcate Services.

SUMMARY:
The purpose of the study is to determent whether there is a difference between two types of treatments in physiotherapy (individual vs group) for patients with low back pain (LBP), in terms of their sensation of how they have been helped and their treatments' outcomes measures. The study hypothesizes are: a) Based on the results of literature review which does not reveal a clear difference between group and individual treatments' outcomes for LBP, it is hypothesized that no difference will be found in treatment results for the two types of group treatments in the present study also, b) The assumption is that different distribution of therapeutic factors will be found in the two types of treatments (individual, group), C) Patients' sensation of how they have been helped will be connected to treatment results.

DETAILED DESCRIPTION:
200 patients with LBP looking for physiotherapy treatment in 15 clinics at Maccabi Healthcare Service in Israel will be recruited. (100 after competion individual therapy, 100 after competion of group therapy). As part of the regular routine in these clinics, patients will be asked to fill the LFSQ, a questionnaire which deals with their back functional status, their level of pain and fear avoidance of physical activity before and after treatment. In the present study, patients will be asked to fill the LFSQ again, 6 months after treatment completion. In two weeks from treatment completion, patients will be interviewed on the telephone. The interview will focuse on their sensation of how they have been helped. It will include an open-ended question and 18 closed questions.

The main study variables will include: participants' perception of functional status, level pain, level of fear avoidance of physical activity, patient-therapist bonding, and helpful therapeutic impacts (client's sense of how she or he has been helped).

ELIGIBILITY:
Inclusion Criteria:

* Low back pain,
* 18 years old and older
* Hebrew speakers , who filled the LFSQ (Lumbar Functional Status Questionnaire) at first visit
* Agreed to participate in this study

Exclusion Criteria:

* Pregnant
* After back or hip operation in the last year
* Back problem from non- orthopedic origin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults (18 years old and older) seeking for physiotherpy treatment for low back pain in one of the 15 clinics participating in this study
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
lumbar functional status | at first and last visit and after 6 months
  participants are asked to fill the LFSQ - lumbar functional status questionnaire before and after tretment completion and after 6 months

SECONDARY OUTCOMES:
patients' perception on how they have been helped | in two weeks after the last visit
  data for this outcome measure will be collected through a telephone interview

OTHER OUTCOMES:
level of pain = NRPS | before and after treatment and after 6 months
  self perception of patients' level of pain will be collected through the NRPSQ=numeric rate pain scale questionnaire
fear avoidance beliefs = FABS | before and after last treatment and after 6 months
  FABS Questionnaire will be used to assess the level of fear of physical activity

CONTACTS AND LOCATIONS:
Overall Officials: Marina Sigal, MD, Principal Investigator — Maccabi Health Service
Locations (1):
- Maccabi Healthcare Services, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: Undecided